CLINICAL TRIAL: NCT06400186
Title: Movement Amplification Gait Training to Enhance Walking Balance Post-Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B4882-P; 1I21RX004882 (NIH)
Record Dates: First submitted 2024-04-26; First posted 2024-05-06 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Chronic Hemiparetic Stroke
Keywords: gait; balance; walking; locomotion; stroke; rehabilitation robotics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biomechanical Response to Balance Challenging Environments (Experimental): Aim 1 will determine how people with chronic stroke (PwCS) adapt their gait in response to different balance challenging environments. For Aim 1, the investigators will conduct a single-session cross sectional study to assess gait patterns during and immediately following walking practiced in balance challenging environments. PwCS will perform treadmill walking in a natural unmodified environment, and in two balance-challenging environments that will include a Movement Amplification Environment (MAE), and an unpredictable lateral perturbation environment. All enrolled participants will undergo clinical outcome measure assessments to identify baseline function. In addition, all participants in Aim 1 will undergo biomechanical testing while walking in each of the three environments to assess changes in their walking patterns.
  Interventions: Behavioral: Treadmill walking in varying external environments
- Heart Rate Response to Balance Challenging Environments (Experimental): Aim 2 is a feasibility study to determine if high intensity gait training can be achieved within a MAE. For Aim 2, the investigators will employ a two-way cross over study design consisting of two gait training sessions (one in a natural unmodified environment and the other in a MAE). The investigators will examine cardiovascular response, perceived exertion, and gait characteristics (speed, number of steps) to quantify if the MAE impacts training intensity. All enrolled participants will undergo clinical outcome measure assessments. In addition, all participants for Aim 2, heart rate (HR), rate of perceived exertion (RPE), number of steps taken during the training sessions, and walking speeds will be recorded.
  Interventions: Behavioral: High intensity gait training in varying external environments

INTERVENTIONS:
Behavioral: High intensity gait training in varying external environments — Participants will engage in two 45-minutes treadmill-based gait training sessions. These training sessions will occur on separate days. One session will be performed in a natural unmodified environment. One session will be performed in a movement amplification environment. The goal of each session will be to achieve 40-minutes of walking within a target heart rate range of 70-85% of estimated heart rate max. Each session will begin and end with a 2.5 minute warm-up and cool down respectively. Participants will be given rest breaks as needed.
  Arms: Heart Rate Response to Balance Challenging Environments
Behavioral: Treadmill walking in varying external environments — Participants will perform a series of treadmill walking trials. Each trial will consist of 400 total steps. The first 100 steps will be performed in a natural unmodified environment. The next 200 steps will be performed in 1 of 3 external environments (natural unmodified, movement amplification, or unpredictable lateral perturbations). The final 100 steps will be performed in a natural unmodified environment. Participants will be given rest breaks between trials.
  Arms: Biomechanical Response to Balance Challenging Environments

SUMMARY:
Stroke is a leading cause of disability in the United States, affecting approximately 795,000 people annually. The Veteran's Health Administration provides over 60,000 outpatient visits for stroke-related care annually at a cost of over $250 million. Among ambulatory people with chronic stroke (PwCS), impaired balance is a common health concern that substantially limits mobility (those with the worst balance walk the least). This project will explore adaptive strategies employed by PwCS in balance challenging environments and if a novel gait training intervention using a robotic device to amplify a person's self-generated movements can improve walking balance. The development of effective interventions to increase walking balance among PwCS will positively impact Veterans' health, quality of life, and ability to participate in walking activities.

DETAILED DESCRIPTION:
Background: There is a pressing need to develop effective methods to enhance walking balance in people with chronic stroke (PwCS). Interventions that amplify self-generated movements may accelerate motor learning by enhancing a person's perception of movement errors. This method could potentially be applied to help PwCS improve walking balance. To this end, the investigators have developed a cable-driven robot to create a Movement Amplification Environment (MAE) during treadmill walking. The MAE challenges walking balance by applying lateral forces to the pelvis that are proportional in magnitude to real-time lateral center of mass (COM) velocity.

Unlike a popular form of balance training that uses unpredictable perturbations to enhance reactive balance, training in a MAE targets anticipatory balance by developing predictive control mechanisms that are likely to persist when the training environment is removed (after-effects). The investigators believe that supplementing high-intensity gait training (the recommended practice to improve walking speed and distance) with a MAE will substantially enhance walking balance. Thus, the purpose is to evaluate the unique effects of MAE training on walking balance in PwCS and determine feasibility of conducting high-intensity gait training in a MAE.

Specific Aims: Aim 1: To evaluate gait patterns PwCS adapt during and immediately following walking practiced in two balance-challenging training environments: MAE and unpredictable lateral perturbations. Aim 2: To establish feasibility of high intensity gait training in MAE the investigators will evaluate cardiovascular intensity during gait training interventions performed in either a natural unmodified environment or a MAE.

Approach: Aims 1: 15 PwCS will participate in a single-day experiment evaluating gait biomechanics (COM dynamics and stepping patterns) during and immediately following treadmill walking performed in a MAE or while receiving frequent unpredictable lateral perturbations. Outcomes will assess if changes in gait patterns to maintain stability persist immediately following exposure to either of the balance-challenging environments. Aim 2: 15 PwCS will participate in two high-intensity gait training sessions. One session will be performed in a natural unmodified environment, the other in a MAE. The investigators will quantify differences in mean heart rate (HR) between the two sessions and whether mean HR is in the target high-intensity range of 70-85% of maximum HR.

Impact: This project will identify if and how PwCS uniquely adapt locomotor strategies following exposure to balance challenging environments and evaluate feasibility of administering high-intensity gait training in a MAE. Training walking balance of PwCS in a MAE by amplifying their own self-generated movements is a radical departure from current practice and could substantially enhance walking balance. Successful outcomes will motivate a future randomized controlled trial assessing the efficacy of MAE training to enhance walking balance in PwCS.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic stroke (more than 6 months post-stroke) with weakness on one side
* Ability to ambulate over ground for 10 meters with or without a single cane, and/or ankle-foot orthosis
* Ability to tolerate 10 minutes of standing

Exclusion Criteria:

* Presence of cognitive impairment (score of 22/30 on the Montreal Cognitive Assessment scale (MoCA))
* Presence of aphasia (score of 71/100 on the Mississippi Aphasia Screening Test (MAST))
* Excessive spasticity in lower limbs (score of > 3 on the Modified Ashworth Scale
* Severe cardiovascular and pulmonary disease affecting gait and balance
* History of recurrent fractures or known orthopedic problems in the lower extremities (i.e. heterotopic ossification) affecting gait and balance
* Concomitant central or peripheral neurological injury (i.e. traumatic head injury or peripheral nerve damage in lower limbs) affecting gait and balance
* Evidence of cerebellar ataxia
* Presence of unhealed decubiti or other skin compromise
* Enrollment in concurrent physical therapy or research involving gait or balance training
* Use of braces/orthotics crossing the knee joint
* Known pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Lateral center of mass (COM) excursion during walking | Arm 1 only: On Day 1 of the study, participants will perform three 5-minute treadmill walking trials. We will measure Lateral COM excursion every gait cycle during each trial.
  Lateral COM excursion is the peak-to-peak distance the COM moves from side-to-side during a complete gait cycle. This distance is measured in meters. Smaller values indicate better ability to control motion during walking.
Minimum lateral margin of stability | Arm 1 only: On Day 1 of the study, participants will perform three 5-minute treadmill walking trials. We will measure minimum lateral margin of stability every gait cycle during each trial.
  Minimum lateral margin of stability is the smallest distance between the lateral extrapolated center of mass position (XCOM) and the lateral base of support (BOS), approximated as the lateral position of the 5th metatarsal marker on the side of the last initial contact. Minimum MOS is identified during stance phase of each step. Extrapolated center of mass (XCOM) position is calculated using:
  XCOM= COM + COM* l/g The minimum lateral margin of stability is calculated in meters. Smaller values indicate greater ability to control motion during walking.
Heart Rate | Arm 2 only: On Day 1, participants will perform 45 minutes of treadmill walking. Seven days later, participants will perform another 45 minutes of continuous treadmill walking. We will measure average HR during every 3-minutes of treadmill walking.
  Participants heart rate in beats per minute (bpm) will be collected to determine cardiovascular response to exercise. Larger heart rates will indicate a stronger cardiovascular response to exercise.
Perceived Exertion (RPE) | Arm 2 only: On Day 1, participants will perform 45 minutes of treadmill walking. Seven days later, participants will perform another 45 minutes of continuous treadmill walking. We will measure average RPE during every 3-minutes of treadmill walking
  Participants exertion monitored via 6-20 point rate of perceived exertion scale and heart rate will be collected to determine participants performance during each training session and track their progress. Minimum score for perceived exertion is 6 and maximum score is 20. Higher score indicates greater exertion and lower score indicates less exertion.
Treadmill walking speed | Arm 2 only: On Day 1, participants will perform 45 minutes of treadmill walking. Seven days later, participants will perform another 45 minutes of continuous treadmill walking. We will measure average speed during every 3-minutes of treadmill walking
  Treadmill speed is a measure of how fast a person is walking on a treadmill. This measure is in units of meters/second. Higher values indicate faster walking speeds.
Number of Steps | Arm 2 only: On Day 1, participants will perform 45 minutes of treadmill walking. Seven days later, participants will perform another 45 minutes of continuous treadmill walking. We will measure the total number of steps during each day.
  An activity monitor worn on the ankle during treadmill walking will identify and record each time a person takes a step. A higher number will indicate a greater number of steps were taken.

SECONDARY OUTCOMES:
Step Length | Arm 1 only: On Day 1 of the study, participants will perform three 5-minute treadmill walking trials. We will measure step length every gait cycle during each trial.
  Step length is calculated as the fore-aft distance between the calcanei markers at initial foot contact. This distance is measured in meters. Larger values indicate longer steps.
Step Width | Arm 1 only: On Day 1 of the study, participants will perform three 5-minute treadmill walking trials. We will measure step width every gait cycle during each trial.
  Step width is calculated as the medio-lateral distance between the left and right 5th Metatarsal markers at initial foot contact. This value is measured in meters. Larger values indicate a wider step.
10 Meter Walk Test (10MWT) | The 10MWT will be administered one time only. This test will be administered on Day 1 before the study intervention has been administered.
  10MWT is a simple measurement of an individual's average walking speed measured at self-selected speed (instruction: "walk at your normal comfortable pace") and fastest-possible speed (instruction: "as fast as you safely can").
Timed Up and Go (TUG) | The TUG will be administered one time only. This test will be administered on Day 1 before the study intervention has been administered.
  TUG is used to assess functional mobility, walking balance, and fall risk. It is a quick, valid, reliable and widely used clinical performance based measure in individuals post-stroke. While there is no time limit to the TUG test, more time taken to finish the task indicates poor balance and greater fall-risk.
Berg Balance Scale (BBS) | The BBS will be administered one time only. This test will be administered on Day 1 before the study intervention has been administered
  BBS is a 14-item measure that assesses static balance with excellent validity and reliability in individuals post-stroke. The total score for this test is 56. Minimum score is 0 and maximum score is 56. Higher scores indicate better balance and lower fall-risk, while lower scores indicate poor balance and increased fall-risk.
Activities-specific Balance Confidence (ABC) Scale | The ABC will be administered one time only. This test will be administered on Day 1 before the study intervention has been administered.
  ABC scale is a self-reported measure of an individual's confidence while performing specific postural and ambulatory activities. The ABC is a reliable and valid measure of balance confidence in individuals post-stroke. The total score for ABC scale is 1600. Minimum score is 0 and maximum score is 1600. Higher scores indicate better balance confidence, while lower scores indicate poor balance confidence
Dynamic Gait Index (DGI) | The DGI will be administered one time only. This test will be administered on Day 1 before the study intervention has been administered.
  DGI is an eight item test that assesses gait, balance and fall risk during usual steady-state walking and walking during more challenging tasks. The total score for this test is 24. Minimum score is 0 and maximum score is 24. Higher scores indicate better walking balance, while lower scores indicate poor walking balance.
Chedoke-McMaster Stroke Assessment (CMSA) scale | The CMSA will be administered one time only. This test will be administered on Day 1 before the study intervention has been administered.
  CMSA will be collected to determine the level of stroke impairment in participants leg and foot. Each domain (leg and foot) are scored on a 7-point scale (stage 1 through 7, most impairment through to no impairment, respectively). Minimum score is 0 and maximum score is 7

CONTACTS AND LOCATIONS:
Overall Officials: Keith Edward Gordon, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois

IPD SHARING:
Plan to Share IPD: Yes
The investigators will create and share de-identified, anonymized data sets. Data sets will be open file formats that include documentation of the material. The investigators will link data sets to associated study publications. Final data sets will be made available as per Hines VA Hospital local policy for long term storage and access until enterprise-level resources become available. These data will be available upon request by researchers and scientists in accordance with federal guidelines and Hines local policy.
  The final data sets will be sufficient for anyone to perform analogous or supplemental analyses that would permit validation of the analysis and results.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available following the completion and publication of study results.
Access Criteria: Data will be publicly available.